CLINICAL TRIAL: NCT03324516
Title: The Effect of Temporal Muscle Suspension of Temporal Hollowing: A Prospective Randomized Clinical Trial
Brief Title: The Effect of Temporal Muscle Suspension of Temporal Hollowing
Acronym: TMS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to limited support staff and time, study was unable to get started
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00120812
Record Dates: First submitted 2017-10-19; First posted 2017-10-27 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Temporal Wasting
Keywords: pterional incision; Temporal hollowing

STUDY DESIGN:
Masking Description: Patients will be given assigned a research limb the morning of the surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients included in this arm will undergo a traditional bony pterional approach for their craniotomy. A superior cuff of temporal muscle will be left attached to the temporal bone.
  Interventions: Procedure: Re-Suspension of the temporal muscle after a craniotomy.
- Control (Active Comparator): Patients included into this arm will receive a traditional pterional approach for their craniotomy. The temporal muscle will be detached in its entirety.
  Interventions: Procedure: Traditional re-suspension of the temporal muscle

INTERVENTIONS:
Procedure: Re-Suspension of the temporal muscle after a craniotomy. — The temporal muscle cuff will be used to re-suspend the temporal muscle after a traditional craniotomy.
  Arms: Experimental Group
Procedure: Traditional re-suspension of the temporal muscle — The temporal muscle will be re-suspended to the bone plate that is used to fixate the temporal bone that is removed for the craniotomy.
  Arms: Control

SUMMARY:
The primary objective is to identify which patients undergoing a traditional pterional approach with 2 different surgical techniques for TMS (Temporal Muscle Suspension) will develop TH (Temporal Hollowing. Pre and post-operative CT scans will be reviewed and analysis with previously proven metrics will be performed.

DETAILED DESCRIPTION:
The pterional approach is an indicated neurosurgical approach commonly used for anterior circular aneurysms, suprasellar lesions, and medial sphenoid wing tumors (1,2). A curvilinear incision from the midline widows peak and extending laterally to 1 cm anterior to the tragus of the ear, terminating within a skin crease, with preservation of the superficial temporal artery if possible. The temporalis fascia is encountered and divided. Either the entire temporalis muscle can be elevated or a cuff of temporalis muscle can be left on the cranium to facilitate closure and suspend the temporalis muscle. Subperiosteal dissection of the muscle is performed and the craniotomies are then accomplished.

Reconstruction of the pterional approach can be accomplished with bony fixation of the bone flap. However, the TMS can be performed by:

1. Resuspension of the temporalis muscle to the cuff of muscle left on the temporal crest or
2. Suturing the temporalis muscle directly to one of the bone plates that is used to for fixation.

The purpose of this prospective study is see if traditional techniques to the closure and temporal muscle suspension (TMS) after the pterional approach will show any differences in post-operative temporal hollowing (TH).

ELIGIBILITY:
Inclusion Criteria:

* This study will include all patients over the age of 18 years who qualify for a pterional approach for their neurosurgical pathology.

Exclusion Criteria:

* Excluded patients will be protected populations, such as inmates or children. Patients will not be excluded on the basis of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in temporal hallowing | 12 months
  The primary end point and outcome variable will the CT quantitative evaluation of temporal hollowing. Percent change and volume analysis as compared to the non operated temporal region in a two dimensional and three dimensional view in a CT Scan of the head and face will be the primary outcome variable.

SECONDARY OUTCOMES:
Patient satisfaction for aesthetic results | 12 months
  Patients will be asked to rate their satisfaction of their aesthetic result on a scale from 1 to 10 with 1 being No satisfaction and 10 being complete satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Gordon, DO, Principal Investigator — Johns Hopkins Department of Plastics and Reconstructive Surgery
Locations (1):
- Johns Hopkins Outpatient CENTER, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Badie B. Cosmetic reconstruction of temporal defect following pterional [corrected] craniotomy. Surg Neurol. 1996 Apr;45(4):383-4. doi: 10.1016/0090-3019(95)00452-1. PMID 8607091
- [Background] Figueiredo EG, Deshmukh P, Nakaji P, Crusius MU, Crawford N, Spetzler RF, Preul MC. The minipterional craniotomy: technical description and anatomic assessment. Neurosurgery. 2007 Nov;61(5 Suppl 2):256-64; discussion 264-5. doi: 10.1227/01.neu.0000303978.11752.45. PMID 18091240

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03324516/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03324516/ICF_001.pdf